CLINICAL TRIAL: NCT03662529
Title: Neurobehavioral Measurement of Substance Users in an Outpatient Treatment Setting
Brief Title: Neurobehavioral Measurement of Substance Users in Outpatient Treatment Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hunter Holmes Mcguire Veteran Affairs Medical Center (U.S. Federal Agency)
Collaborators: VA Mental Illness Research, Education and Clinical Centers (U.S. Federal Agency)
Responsible Party: Principal Investigator, James Bjork, Neuroscientist, Hunter Holmes Mcguire Veteran Affairs Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 02287
Record Dates: First submitted 2018-08-17; First posted 2018-09-07 (Actual); Last update posted 2018-09-07 (Actual); Status verified 2018-09

CONDITIONS: Cocaine Dependence; Cocaine Use Disorder; Opiate Dependence; Opioid-use Disorder; Cannabis Dependence
MeSH Terms: conditions — Cocaine-Related Disorders; Opioid-Related Disorders; Marijuana Abuse | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Participants were effectively block-randomized either into individual treatment as usual (TAU)(practitioners who administered TAU) OR individual therapy with the study intervention (Mind Freedom Plan), where data from both arms was collected in parallel.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mind Freedom Plan therapy sessions (Experimental): The Four-Session Mind Freedom Plan (MFP) is cognitive behavioral therapy (CBT)-based, client-centered, manualized individual therapy that functions as part of intensive outpatient substance abuse treatment. The MFP model is based on efficacious brief interventions, with content and format driven from military veteran feedback. The four 60-minute MFP sessions were one-on-one private consultations with a therapist that were focused on identifying and changing unhealthy thinking and behavioral patterns as core elements of CBT, but with an emphasis on problem-solving, coping skills, goal setting, and psychosocial functioning. At each session, structured worksheets were utilized and homework was assigned to facilitate this CBT-based skill building.
  Interventions: Behavioral: Four-Session Mind Freedom Plan
- Treatment as usual therapy (Active Comparator): The four 50-minute TAU sessions were one-on-one individual therapy sessions. Therapy was mostly supportive therapy with an emphasis problem solving on increasing veteran motivation. A discussion of the antecedents to relapse would take place if a relapse occurred and coping skills were discussed and reviewed. Veterans were also connected with community-level psychosocial supports as appropriate.
  Interventions: Behavioral: Treatment as usual therapy

INTERVENTIONS:
Behavioral: Four-Session Mind Freedom Plan — Problem-solving-focused individualized cognitive behavioral therapy (CBT) that featured homework-worksheets to reinforce session-concepts.
  Other Names: Mind Freedom Plan
  Arms: Mind Freedom Plan therapy sessions
Behavioral: Treatment as usual therapy — Therapy was mostly supportive therapy with an emphasis problem solving on increasing veteran motivation. A discussion of the antecedents to relapse would take place if a relapse occurred and coping skills were discussed and reviewed.
  Other Names: Treatment as usual
  Arms: Treatment as usual therapy

SUMMARY:
This study was an internal program effectiveness evaluation of the effects of a four-session weekly individualized cognitive therapy program (called the "Mind Freedom Plan" (MFP)) on substance use outcomes and substance abuse treatment retention in Veterans admitted to an intensive outpatient treatment program for substance abuse at the Richmond Veterans Administration Medical Center (RICVAMC). Substance use and treatment retention metrics of MFP-assigned Veterans were compared with those of Veterans assigned to typical case-management-oriented weekly individual sessions.

DETAILED DESCRIPTION:
This study was funded and launched as an internal program evaluation regarding the effects of a four-session weekly individualized cognitive therapy program called the "Mind Freedom Plan" (MFP) on substance use outcomes, impulsivity, and substance abuse treatment retention in veterans admitted to the intensive outpatient (treatment) program (IOP) for substance abuse at the Richmond Virginia Hunter Holmes McGuire Veterans Administration Medical Center (RICVAMC). Substance use and treatment retention outcomes were compared between veterans randomly assigned to the MFP versus treatment as usual (TAU), which consisted of typical case-management-oriented weekly individual sessions. Veteran participants were approached and consented within a week of admission to the RICVAMC IOP and randomly assigned to either an MFP or TAU practitioner. Assignment was constrained by practitioner new-patient availability in order to place veterans into individualized care sessions as soon as possible.

Participants completed self-reported and interview-based mood, personality and addiction severity assessments at study entry. After one month, participants were reassessed with psychometric symptomatology questionnaires, and also completed a 60-minute neurobehavioral testing session in a follow-up appointment. Subjects completed the Delis-Kaplan Executive Function System (DKEFS) Tower Test of planning ability, along with a delay-discounting decision-making task, a stop-signal task, and a go-nogo behavior inhibition task that used emotional and expressionless faces as stimuli.

ELIGIBILITY:
Inclusion Criteria:

* Enrollment in the Substance Abuse Treatment Program - Intensive Outpatient Program
* Currently meets criteria for an Alcohol or Substance Use Disorder per SUD clinic intake

Exclusion Criteria:

* Unable to read and speak English
* Currently active-duty military
* Current engaged with legal involvement that is mandating the completion of the substance use program.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2017-06-05 (Actual); Primary Completion 2018-01-08 (Actual); Study Completion 2018-02-01 (Actual)

PRIMARY OUTCOMES:
Percent of patients who completed the Substance Abuse Treatment Program (SATP) Intensive Outpatient Program (IOP). | 28-Day
  Chart review variable; SATP IOP patients are designated as completers vs non-completers by their IOP social worker. IOP treatment retention outcome is documented in the patients' charts as part of standard care.
Rate of abstinence during final week of intensive outpatient therapy (IOP) | 21-28 Days
  Chart review variable; abstinence in the final week of IOP was defined as urine drug screen (UDS) negative and no self-reported substance use by the final week of IOP. UDS results and self-reported substance use are documented in the patients' charts as part of standard care.

SECONDARY OUTCOMES:
Drug use during outpatient therapy | 1-28 Days
  Proportion of drug-negative urine samples during 4-week outpatient treatment
Decision-based impulsivity | 28 Days
  Severity of delay-discounting behavior in laboratory task
Rapid-response impulsivity | 28 Days
  Stop signal reaction time (SSRT) in stop-signal computer task
Problem-solving ability | 28 Days
  Mean difference in Delis-Kaplan Executive Function System (D-KEFS) Tower Subtest total score at 4-week follow up with MFP vs TAU. The D-KEFS Tower Test is a cognitive test for executive functioning, planning, and problem-solving ability. During the D-KEFS Tower Test, participants are instructed to create towers using discs and a set of pegs that correspond to a model. D-KEFS Tower Test total scores range from 0 to 30, with higher scores indicating a better performance on the tower building task.
Depression symptomatology | Pre-treatment baseline and 28 Days
  Change in Beck Depression Inventory (BDI)-II total scores from baseline to 4-week follow up with MFP vs TAU. Depressive symptom severity was measured with the total score of the 21-item BDI-II. BDI-II total scores range from 0 to 63, with higher scores represent increased depressive symptoms.
Quality of life as assessed by the Quality of Life Inventory (QoLI) total score. | Pre-treatment baseline and 28 Days
  Change in Quality of Life Inventory (QoLI) total scores from baseline to 4-week follow up with MFP vs TAU. The QoLI is a 32-item self-report instrument that assesses positive mental health, wellbeing, and happiness using an overall score across 16 life domains (e.g., health, work). Participants rate how important each domain is (0-2 scale) and how satisfied they are with this area of their life (7-point scale). QoLI satisfaction scores are weighted based on importance rating in order to create a total score.
Impulsive personality | Pre-treatment baseline and 28 Days
  Change in Barratt Impulsiveness Scale (BIS-11) total scores from baseline to 4-week follow up with MFP vs TAU. Total score on the 30-item (4-point scale) BIS-11 is a self-report measure of trait impulsivity, with higher scores reflecting increased impulsivity.

CONTACTS AND LOCATIONS:
Overall Officials: James M Bjork, PhD, Principal Investigator — Hunter Holmes McGuire VA Medical Center
Locations (1):
- Hunter Holmes McGuire VA Medical Center, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2017-06-14): https://cdn.clinicaltrials.gov/large-docs/29/NCT03662529/Prot_000.pdf